CLINICAL TRIAL: NCT04267315
Title: Trigger Point Injections for Post-Mastectomy Pain Syndrome: A Double-Blind Randomized Controlled Trial With Intention-to-Treat Analysis
Brief Title: Trigger Point Injections for Post-Mastectomy Pain Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Collaborators: Hospital de Câncer de Barretos (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1474/19
Record Dates: First submitted 2020-01-29; First posted 2020-02-12 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Post-mastectomy Pain Syndrome; Myofascial Pain Syndrome; Trigger Point Pain, Myofascial; Breast Cancer
MeSH Terms: conditions — Myofascial Pain Syndromes; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Double-blind randomized controlled trial comparing the efficacy of TPI + standard of care (ACTIVE) versus sham TPI + standard of care(PLACEBO), with an intention-to-treat analysis
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patients will be randomized as they enter the study (T0). Only one of the researchers will have access to the randomization list. The researcher responsible for the procedure will receive an email at the day of the first injection, informing of the participant's allocation group. The outcomes assessor, patient, attending Physiatrist and the Rehabilitation team will be blinded to the patient's allocation group until the end of the study. Only the researcher the performed the TPI, and the researcher responsible for the allocation list will have access to that information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): 3 weekly sessions of TPI. Participants will undergo 1mL injections of 1% lidocaine in the muscles identified with either active or latent trigger points at the initial assessment. The same muscles will be injected at all procedures.
  Interventions: Procedure: Trigger point injection; Other: Comprehensive Rehabilitation program
- Placebo (Sham Comparator): 3 weekly sessions of subcutaneous saline injections. Participants will undergo 0.2mL subcutaneous saline injections superficial to the trigger points identified at initial assessment. The same superficial sites will be injected in all procedures.
  Interventions: Procedure: Subcutaneous saline injection; Other: Comprehensive Rehabilitation program

INTERVENTIONS:
Procedure: Trigger point injection — 1mL injections of 1% lidocaine in the muscles identified active trigger points at the day of intervention (pectoralis major, serratus anterior, levator scapulae, latissimus dorsi, infraspinatus).
  Arms: Active
Procedure: Subcutaneous saline injection — 0.2mL subcutaneous saline injections superficial to the muscles identified with active trigger points at the day of intervention (pectoralis major, serratus anterior, levator scapulae, latissimus dorsi, infraspinatus).
  Arms: Placebo
Other: Comprehensive Rehabilitation program — Patients in both groups will undergo standard of care rehabilitation delivered by a Physiatrist, which may include Physical Therapy, Occupational Therapy, Exercise Physiologist, Rehabilitation Nurse, Psychologist, as per Physiatrist's prescription. Both the comprehensive rehabilitation program and pain medications will continue to be managed by participant's Physiatrist, who will be blinded to patient's allocation. The researchers will be responsible for TPI and for data collection.

SUMMARY:
Post-Mastectomy Pain Syndrome (PMPS) is a chronic pain that persists for more than three months after a surgical breast procedure. It has 11-70% incidence in patients that underwent a breast surgery. It consists of mixed pain, frequently associated with myofascial pain, an specific type of muscular pain. Trigger point injections (TPI) are classically used for the treatment of myofascial pain in other painful conditions. However, there are no controlled trials assessing the efficacy of TPI in the treatment of PMPS. The intervention objective is to assess the efficacy of TPI in patients with PMPS, when associated with a comprehensive rehabilitation program and pain management.

DETAILED DESCRIPTION:
INTRODUCTION: Post-Mastectomy Pain Syndrome (PMPS) is a chronic pain that persists for more than three months after a surgical breast procedure. It has 11-70% incidence in patients that underwent a breast surgery. It consists of mixed pain, frequently associated with myofascial pain. Trigger point injections (TPI) are classically used for the treatment of myofascial pain in other etiologies. However, there are no controlled trials assessing the efficacy of TPI in the treatment of PMPS

OBJECTIVE: Assess the efficacy of TPI in patients with PMPS, when associated with a comprehensive rehabilitation program and pain management.

METHODS: Double-blind randomized controlled trial with intention-to-treat analysis. Both groups will undergo standard of care delivered by Physiatrist blinded to group allocation. Active group will undergo TPI with 1% lidocaine in each identified trigger-point, weekly, for three consecutive weeks. Control group will undergo subcutaneous saline injection superficial to the same trigger points, with the same frequency and number of sessions. Primary outcome is the mean difference between groups for pain levels, as assessed by Visual Numeric Scale (VNS), from baseline to 3 months after the procedure.

STATISTICAL ANALYSIS: Difference between groups at baseline, one and three months after injection, using Analysis of Covariance (ANCOVA) for the following outcomes: VNS; Presence of active trigger points, Pressure pain threshold (PPT); Short-Form McGill Pain Questionnaire (SF-MPQ); Neuropathic Pain Symptom Inventory (NPSI); Disabilities of the Arm, Shoulder and Hand Questionnaire (DASH); Range of motion (ROM) of affected shoulder, for abduction and external rotation; adverse events; use of pain medication.

Total sample size is 120. Alpha=5%, power=80%.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients.
* PMPS diagnosis, as per Wisotzky et col.

  * Pain > 3 months over breast, chest wall or shoulder ipsilateral to surgery.
* Pain Visual analog Scale (VAS) ≥4.
* At least one active trigger point in the following muscles: pectoralis major, superior trapezius, serratus anterior, levator scapularis, latissimus dorsi, infraspinatus

Exclusion Criteria:

* Current radiation therapy or time since completion < 3months.
* Allergy to lidocaine or other local anesthetics
* Active infection over injection sites
* Unavailability to be at the hospital during study intervention.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-02-15 (Estimated)

PRIMARY OUTCOMES:
Visual Numeric Scale (VNS) for pain in 3 months | 3 months
  Mean difference of Pain between groups from baseline to 3 months(T3m), assessed by the Visual Numeric Scale (VNS, 0-10), in which higher scores represent higher pain intensity.
Trigger-points | 1 month
  Number of active trigger-points in the assessed muscles (latissimus dorsi, levator scapulae, trapezius superior, infraspinatus, pectoralis major, serratus anterior). Mean difference between groups.
Trigger-points | 3 months
  Number of active trigger-points in the assessed muscles (latissimus dorsi, levator scapulae, trapezius superior, infraspinatus, pectoralis major, serratus anterior). Mean difference between groups.
Pressure Pain Threshold (PPT) | 1 month
  Pressure Pain Threshold (PPT) at bilateral latissimus dorsi, levator scapulae, trapezius superior, infraspinatus, pectoralis major, serratus anterior. Difference from baseline
Pressure Pain Threshold | 3 months
  Pressure Pain Threshold (PPT) at bilateral latissimus dorsi, levator scapulae, trapezius superior, infraspinatus, pectoralis major, serratus anterior. Difference from baseline

SECONDARY OUTCOMES:
Visual Numeric Scale (VNS) for pain in 1 month | 1 month
  Mean difference of Pain between groups from baseline,assessed by the Visual Numeric Scale (VNS, 0-10), in which higher scores represent higher pain intensity.
Short-Form McGill Pain Questionnaire (SF-MPQ) - total score, sensorial and affective scale | 1 month
  Short-Form McGill Pain Questionnaire - total score, sensorial and affective scale. Mean difference between groups from baseline. Higher values represent higher pain intensity
Short-Form McGill Pain Questionnaire (SF-MPQ) - total score, sensorial and affective scale | 3 months
  Short-Form McGill Pain Questionnaire - total score, sensorial and affective scale. Mean difference between groups from baseline. Higher values represent higher pain intensity
Neuropathic Pain Symptom Inventory (NPSI) | 1 month.
  Neuropathic Pain Symptom Inventory . Mean difference between groups from baseline. Higher values represent more symptoms of neuropathic pain.
Neuropathic Pain Symptom Inventory (NPSI) | 3 months
  Neuropathic Pain Symptom Inventory . Mean difference between groups from baseline. Higher values represent more symptoms of neuropathic pain.
Disabilities of the Arm, Shoulder and Hand Questionnaire (DASH) | 1 month
  Disabilities of the Arm, Shoulder and Hand Questionnaire (DASH). Mean difference between groups from baseline. Higher values represent lower functionality.
Disabilities of the Arm, Shoulder and Hand Questionnaire (DASH) | 3 months
  Disabilities of the Arm, Shoulder and Hand Questionnaire (DASH). Mean difference between groups from baseline. Higher values represent lower functionality.
Shoulder range of motion (ROM) | 1 month
  Range of motion (ROM) of affected shoulder, for abduction and external rotation. Mean difference between groups from baseline.
Shoulder range of motion (ROM) | 3 months
  Range of motion (ROM) of affected shoulder, for abduction and external rotation. Mean difference between groups from baseline.
Percentage of patients with at least 30% improvement of pain as per VNS scores (VNS30%) | 1 month
  Percentage of patients with at least 30% improvement of pain as per VAS scores (VAS30%). Mean difference between groups.
Percentage of patients with at least 30% improvement of pain as per VNS scores (VNS30%) | 3 months
  Percentage of patients with at least 30% improvement of pain as per VAS scores (VAS30%). Mean difference between groups.
Percentage of patients with at least 50% improvement of pain as per VNS scores (VNS50%) | 1 month
  Percentage of patients with at least 50% improvement of pain as per VAS scores (VAS30%). Mean difference between groups.
Percentage of patients with at least 50% improvement of pain as per VNS scores (VNS50%) | 3 months
  Percentage of patients with at least 50% improvement of pain as per VAS scores (VAS30%). Mean difference between groups.
Adverse events | 1 month
  Number of participants with adverse events. Mean difference between groups.
Adverse events | 3 months
  Number of participants with adverse events. Mean difference between groups.
Pain medication | 1 months
  Use of pain medication. Classified as "Increased", "Decreased", "Stable" or "Non-applicable" . Mean difference between groups.
Pain medication | 3 months
  Use of pain medication. Classified as "Increased", "Decreased", "Stable" or "Non-applicable" . Mean difference between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Christina May Moran de Brito, MD, PhD, Study Director — Instituto do Câncer do Estado de São Paulo
Locations (2):
- Brazil (2):
  - Hospital de Câncer de Barretos, Barretos, São Paulo
  - Instituto do Câncer do Estado de São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wisotzky E, Hanrahan N, Lione TP, Maltser S. Deconstructing Postmastectomy Syndrome: Implications for Physiatric Management. Phys Med Rehabil Clin N Am. 2017 Feb;28(1):153-169. doi: 10.1016/j.pmr.2016.09.003. PMID 27912994